CLINICAL TRIAL: NCT06550544
Title: Hysteroscopic Guided Versus Ultrasound Guided Extraction of Retained IUD A Randomized Controlled Study
Brief Title: Hysteroscopic Guided Versus Ultrasound Guided Extraction of Retained IUD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Bedaya Hospital (Other)
Responsible Party: Principal Investigator, Usama M Fouda, Prof., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Retained IUD/Hysteroscopy/US
Record Dates: First submitted 2024-04-11; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Contraceptive Device; Complications
Keywords: IUD; Office hysteroscopy; Ultrasound; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Office hysteroscopy (Active Comparator): A rigid 2.9 mm hysteroscope with 30° forward oblique lens and outer sheath diameter of 5 mm will be used in the procedure. Vaginoscopic approach will be used. A 5 F grasper will be used to grasp and extract the IUD.
  .Pain intensity will be assessed by visual analogue scale immediately after the procedure.
  Interventions: Procedure: Office hysteroscopy
- Ultrasound guided (Active Comparator): An alligator forceps will be introduced into the uterine cavity under ultrasound sound guidance. The IUD will be grasped and extracted outside the uterus.
  .Pain intensity will be assessed by visual analogue scale immediately after the procedure.
  Interventions: Procedure: Ultrasound guided

INTERVENTIONS:
Procedure: Office hysteroscopy — A rigid 2.9 mm hysteroscope with 30° forward oblique lens and outer sheath diameter of 5 mm will be used in the procedure. Vaginoscopic approach will be used. A 5 F grasper will be used to grasp and extract the IUD.
  Pain intensity will be assessed by visual analogue scale immediately after the procedure.
  Arms: Office hysteroscopy
Procedure: Ultrasound guided — An alligator forceps will be introduced into the uterine cavity under ultrasound sound guidance. The IUD will be grasped and extracted outside the uterus.
  Pain intensity will be assessed by visual analogue scale immediately after the procedure.
  Arms: Ultrasound guided

SUMMARY:
The aim of this randomized controlled study is to compare the pain experienced during extraction of retained IUD by office hysteroscopy with the pain experienced during extraction of retained IUD under ultrasound guidance . Moreover, the success of both procedures was compared. Various subgroups (patients who delivered only by Caesarean section, patients who delivered virginally, nulliparous women and menopausal patients) in both groups are compared.

DETAILED DESCRIPTION:
The intrauterine device (IUD) is a commonly used long-acting, effective and reversible method of contraception. The recommended way to remove a IUD is by grasping the threads with forceps and applying gentle traction until the IUD is extracted from the external os.

Absent of the threads at the time of IUD removal is reported in 4.5 to 18% of cases. If the IUD is present in the uterus and threads are not visible , its removal in the office setting can still be achieved in about 80% of patients with the use of alligator forceps or string retrieval devices, hooks or clamps. However, blind manipulation may cause uterine perforation . In cases where such devices have failed (retained IUD ), If in office extraction of IUD by these instruments failed, removal of this retained IUD in the operating room is often employed because cervical dilatation and regional or general anesthesia are needed.

In the last decade, several studies reported in office extraction of retained IUD by office hysteroscopy or under ultrasound guidance. No studies compared the efficacy or safety of these procedures

ELIGIBILITY:
Inclusion Criteria:

* Patients with retained IUD

Exclusion Criteria:

* Active pelvic infection
* Viable intrauterine pregnancy
* Cervical pathology

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-08-21 (Estimated); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-02-21 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | Immediately after the procedure
  Measured after the procedure using a 10 cm Visual analogue scale ( where 0 indicates no pain') and 10 indicates a 'pain as bad as it could possibly be')

SECONDARY OUTCOMES:
Success of IUD extraction | Immediately after the procedure
  Percentage of successfully extracted IUD (number of extracted IUDs / total number of retained IUDs)

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, Prof., Principal Investigator — Cairo University
Locations (1):
- Obstetrics &Gynecology Department , Faculty of medicine ,Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Townsend L, Luxford E, Mizia K. Effectiveness of ultrasound-guided removal of intrauterine devices. Aust N Z J Obstet Gynaecol. 2022 Oct;62(5):800-802. doi: 10.1111/ajo.13584. Epub 2022 Jul 11. PMID 35815357